CLINICAL TRIAL: NCT03959111
Title: Auricular Acupuncture Stimulation for Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016P000678
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ear stimulation (Location 1) (Experimental)
  Interventions: Other: Stimulation at Location 1
- Ear stimulation (Location 2) (Experimental)
  Interventions: Other: Stimulation at Location 2

INTERVENTIONS:
Other: Stimulation at Location 1 — Stimulation parameters will include 1) density wave adjusted to 20Hz with less than 1 ms pulse width, 2) intensity adjusted based on the tolerance of the patient (moderate tolerable stimulation without pain), and 3) treatment will be applied 1 time per day, 5 times per week for four weeks (on-site tVNS treatment plus self-administration at home).
  Arms: Ear stimulation (Location 1)
Other: Stimulation at Location 2 — Stimulation parameters will include 1) density wave adjusted to 20Hz with less than 1 ms pulse width, 2) intensity adjusted based on the tolerance of the patient (moderate tolerable stimulation without pain), and 3) treatment will be applied 1 time per day, 5 times per week for four weeks (on-site tVNS treatment plus self-administration at home).
  Arms: Ear stimulation (Location 2)

SUMMARY:
This proposal aims to investigate the treatment effect and underlying mechanism of transcutaneous acupuncture stimulation on chronic low back pain. We believe that this study, if successful, will provide new treatment options for chronic low back pain, reduce the use of opioid analgesics in chronic pain management, and enhance our understanding of the underlying mechanism of nerve stimulation treatment, as well as the pathophysiology and development of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers 18-65 years of age.
* Meet the Classification Criteria of chronic LBP (having low back pain for more than 6 months), as determined by a referring physician.
* Received stable treatment or no treatment in the past month.
* At least a 10th grade English-reading level. English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Specific causes of back pain (e.g., epidural abscess, compression fracture, spondyloarthropathy, malignancy, cauda equina syndrome) or radicular pain, radiculopathy, or spinal canal stenosis. Complicated back problems (e.g., prior back surgery, medico-legal issues).
* Presence of headache/migraine, as well as widespread body pain such as fibromyalgia.
* The intent to undergo surgery during participation in the study.
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcomes (e.g., asthma or claustrophobia).
* Presence of any contraindications to MRI scanning (e.g., cardiac pacemaker, metal implants, fear of enclosed spaces, pregnancy, cannot lie still in fMRI scanner).
* Conditions that might confound longitudinal effects or interpretation of results (e.g. severe fibromyalgia, rheumatoid arthritis).
* Pregnant or lactating.
* Conditions making study participation difficult (e.g., paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator during Session 1).
* Active substance abuse disorders within the last 24 months (based on subject self-report).
* Use of prescription steroids for pain during the past six months.
* Presence of any other acute or chronic pain disorder.
* Any medical conditions, such as peripheral neuropathy, that could affect the results of QST.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Low Back Pain Intensity | 4 months
  This is a uni-dimensional measure of pain intensity. It uses an 11-point numeric scale. We will use it to measure the patient's average pain intensity in the past week, which will be measured at the beginning and end of the study.

SECONDARY OUTCOMES:
Roland-Morris Disability Questionnaire score | 4 months
  The modified RMDQ is a self-administered disability measure in cLBP patients.
Patient-Reported Outcomes Measurement Information System (PROMIS) scores | 4 months
  The PROMIS, funded by the NIH, is a system containing reliable, flexible, precise, and responsive assessment tools that have been widely validated in numerous samples. We will use PROMIS-29 to assess pain interferences and intensity, physical function, depression, anxiety, fatigue, and sleep in the past 7 days.
Pain medication dose changes | 4 months
  Pain medication dose changes as determined by a weekly-collected medication log
Pain Catastrophizing Scale | 4 months
  The PCS is a 15-item questionnaire used to characterize an individual's tendency to magnify the threat value of a pain experience and to feel helpless in the presence of pain.
The Pennebaker Inventory of Limbic Languidness | 4 months
  PILL allows individuals to rate how frequently they have experienced each of 54 common symptoms over an unspecified time period in the past using a five-point Likert scale. The PILL contains a range of physical symptoms, including some items that are pain-related (e.g., headache, back pains, sore muscles).

OTHER OUTCOMES:
Resting state functional connectivity changes of the PAG | 1 month
  Functional connectivity changes of the periaqueductal gray while at rest.
Resting state functional connectivity of the medial and lateral hypothalamus | 1 month
  Functional connectivity changes of the hypothalamus while at rest.
CBF as measured by ASL | 1 month
  Changes in cerebral blood flow.
Inflammation biomarkers | 1 month
  Changes in inflammatory biomarker levels

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Li T, Yan K, Wu J, Reddy S, Sacca V, Ursitti AK, Zhu M, Hodges S, Chen L, Kong J. Both Transcutaneous Auricular Vagus Nerve Stimulation and Great Auricular Nerve Stimulation Modulate Functional and Structural Connectivity of Brainstem Nuclei in Chronic Low Back Pain. Neuromodulation. 2025 Oct 15:S1094-7159(25)01025-6. doi: 10.1016/j.neurom.2025.08.415. Online ahead of print. PMID 41091086